CLINICAL TRIAL: NCT00887237
Title: Triple Site Ventricular Stimulation for CRT Candidates
Brief Title: Triple Site Ventricular Stimulation for Cardiac Resynchronization Therapy (CRT) Candidates
Acronym: TRIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIV
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Heart Failure
Keywords: Heart failure; Cardiac resynchronization; Triple site ventricular pacing
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TRIV (Experimental): Cardiac resynchronization with triple site ventricular stimulation (2 RV leads and 1 LV lead)
  Interventions: Device: CRT with triple site ventricular stimulation
- BIV (Active Comparator): Conventional cardiac resynchronization
  Interventions: Device: Conventional cardiac resynchronization

INTERVENTIONS:
Device: CRT with triple site ventricular stimulation — CRT with triple site ventricular stimulation (2 RV leads and 1 LV lead)
  Arms: TRIV
Device: Conventional cardiac resynchronization — Conventional cardiac resynchronization
  Arms: BIV

SUMMARY:
Despite technological progresses the rate of non-responders to cardiac resynchronization therapy (CRT) remains close to 30%. This inconsistent effect of CRT might be due to incomplete resynchronization as dyssynchrony can persist in 25% to 30% of patients during CRT.

One might hypothesize that stimulating the ventricles at a single site is suboptimal and that stimulating multiple left ventricular (LV) or right ventricular (RV) sites may improve ventricular resynchronization and, consequently, its hemodynamic and clinical effects. First studies have suggested that 1 RV + 2 LV pacing sites configurations increased significantly dP/dt, pulse pressure, LV end-diastolic pressure, and is associated with more LV remodeling and better responder rate compared with pacing a single LV site. First studies with 2 RV+LV pacing sites configuration demonstrated increased dP/dt and cardiac output and a decrease of the cardiac dyssynchrony.

The present pilot trial was designed to examine the 6-month safety of biventricular stimulation with 2 right ventricular (RV) and 1 left ventricular (LV) leads - main objective- and to assess its clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* > 18 years old
* Cardiac resynchronization indication : New York Heart Association (NYHA) Class III/IV & QRS width > 120 ms milliseconds (ms) OR NYHA class II & QRS width > 150 ms
* Sinus rhythm
* First implant procedure

Exclusion Criteria:

* Permanent ventricular tachycardia
* Permanent pacing indication for 3rd degree atrioventricular (AV) block
* Diagnosed or suspected acute myocarditis
* Less than 1 year life expectancy related to a non-cardiovascular disease
* Impossibility to perform follow-up in the investigative center
* Pregnant woman
* Patient which may not cooperate to study procedures as evaluated by investigator
* Legally protected adult patient or patient unable to give an informed consent
* Patient enrolled in an other clinical trial
* Patient which does not benefit from a social protection system
* Renal insufficiency
* Patient registered on a heart transplant waiting list
* Disease and/or health condition which may interfere with study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Safety of triple site CRT compared to conventional CRT | 6 months

SECONDARY OUTCOMES:
Feasibility of triple site CRT | 6 months
Left ventricle remodeling | At 3 and 6 months
LV ejection fraction | At 3 and 6 months
Cardiac dyssynchrony | At 3 and 6 months
Functional status (clinical composite score and NYHA class) | At 3 and 6 months
Exercise capacity (6 minutes hall walk test distance) | At 3 and 6 months
Quality of life | At 3 and 6 months
B-Type Natriuretic Peptide (BNP) level | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Anselme, Pr, Principal Investigator — University Hospital, Rouen
Locations (12):
- France (12):
  - University hospital of Bordeaux, Bordeaux
  - University hospital of Lille, Lille
  - University hospital La Timone, Marseille
  - University hospital of Montpellier, Montpellier
  - University hospital of Nancy, Nancy
  - Nouvelles Cliniques Nantaises, Nantes
  - University hospital of Nantes, Nantes
  - Clinique Bizet, Paris
  - University Hospital of Rennes, Rennes
  - University hospital of Rouen, Rouen
  - Centre Cardiologique du Nord, Saint-Denis
  - Hôpital Saint Louis, La Rochelle, Île-de-France Region

REFERENCES:
- [Derived] Anselme F, Bordachar P, Pasquie JL, Klug D, Leclercq C, Milhem A, Alonso C, Deharo JC, Gras D, Probst V, Piot O, Savoure A. Safety, feasibility, and outcome results of cardiac resynchronization with triple-site ventricular stimulation compared to conventional cardiac resynchronization. Heart Rhythm. 2016 Jan;13(1):183-9. doi: 10.1016/j.hrthm.2015.08.036. Epub 2015 Sep 26. PMID 26325531